CLINICAL TRIAL: NCT01192165
Title: An Open-Label, Phase I/Ib Dose Escalation Study to Assess the Safety and Tolerability of GSK1120212 in Combination With Docetaxel, Erlotinib, Pemetrexed, Pemetrexed + Carboplatin, Pemetrexed + Cisplatin, or Nab-Paclitaxel in Subjects With Advanced Solid Tumors
Brief Title: Safety and Tolerability Study of GSK1120212, a MEK Inhibitor, in Combination With Docetaxel, Erlotinib, Pemetrexed, Pemetrexed + Carboplatin, Pemetrexed + Cisplatin, or Nab-Paclitaxel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 113486; 2012-000257-32 (EudraCT Number)
Record Dates: First submitted 2010-08-30; First posted 2010-08-31 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Cancer
Keywords: Taxotere; Cisplatin; Carboplatin; Trametinib; GSK1120212; Tarceva; KRAS; Pemetrexed; MEK inhibitor; nab-Paclitaxel; Docetaxel; Alimta; Abraxane; Erlotinib
MeSH Terms: conditions — Neoplasms | interventions — trametinib; Docetaxel; Erlotinib Hydrochloride; Pemetrexed; Carboplatin; 130-nm albumin-bound paclitaxel; Cisplatin

ARMS (6):
- Treatment Group 1 (Experimental): Trametinib plus Docetaxel
  Interventions: Drug: Trametinib (GSK1120212); Drug: Docetaxel
- Treatment Group 2 (Experimental): Trametinib plus Erlotinib
  Interventions: Drug: Trametinib (GSK1120212); Drug: Erlotinib
- Treatment Group 3 (Experimental): Trametinib plus Pemetrexed
  Interventions: Drug: Trametinib (GSK1120212); Drug: Pemetrexed
- Treatment Group 4 (Experimental): Trametinib plus Pemetrexed and Carboplatin
  Interventions: Drug: Trametinib (GSK1120212); Drug: Pemetrexed; Drug: Carboplatin
- Treatment Group 5 (Experimental): Trametinib plus nab-Paclitaxel
  Interventions: Drug: Trametinib (GSK1120212); Drug: nab-Paclitaxel
- Treatment Group 6 (Experimental): Trametinib plus Pemetrexed and Cisplatin
  Interventions: Drug: Trametinib (GSK1120212); Drug: Pemetrexed; Drug: Cisplatin

INTERVENTIONS:
Drug: Trametinib (GSK1120212) — Investigational small molecule targeted therapy (MEK1/2 inhibitor)
Drug: Docetaxel — Chemotherapy
  Arms: Treatment Group 1
Drug: Erlotinib — Small molecule targeted therapy (EGFR inhibitor)
  Arms: Treatment Group 2
Drug: Pemetrexed — Chemotherapy
  Arms: Treatment Group 3; Treatment Group 4; Treatment Group 6
Drug: Carboplatin — Chemotherapy
  Arms: Treatment Group 4
Drug: nab-Paclitaxel — Chemotherapy
  Arms: Treatment Group 5
Drug: Cisplatin — Chemotherapy
  Arms: Treatment Group 6

SUMMARY:
The purpose of this study is to determine what dose of GSK1120212 can be given safely in combination with at least one other drug that is already approved to treat cancer. This study will test the safety of up to 6 different GSK1120212 study treatment combinations (GSK1120212 plus either docetaxel, erlotinib, pemetrexed, pemetrexed + carboplatin, pemetrexed + cisplatin, or nab-paclitaxel). The doses identified in this study may be used in future trials to test whether the combination treatment is a safe and effective therapy for subjects with metastatic lung and/or pancreatic cancers.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a solid tumor. Expansion cohorts are limited to non-small cell lung cancer and/or pancreatic cancer with or without a KRAS mutation.
* Tumor progression following at least one prior standard therapy, the subject refuses standard therapy, or no standard therapy exists.
* The subject has a radiographically measurable tumor.
* The subject is able to carry out daily life activities without difficulty.
* The subject is able to swallow and retain oral medication.
* The subject does not have significant side effects from previous anti-cancer treatment.
* The subject has adequate organ and blood cell counts.
* Sexually active subjects must use medically acceptable methods of contraception during the course of the study.

Exclusion Criteria:

* The subject has had major surgery or received certain types of cancer therapy within 2-3 weeks before starting the study.
* The subject has a brain tumor.
* Current severe, uncontrolled systemic disease.
* History of clinically significant heart, lung, or eye/vision problems.
* The subject has high blood pressure that is not well-controlled with medication.
* The subject has a permanent pacemaker.
* The subject is pregnant or breastfeeding.
* Positive for Hepatitis B, Hepatitis C, or HIV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2010-09-14 (Actual); Primary Completion 2013-10-07 (Actual); Study Completion 2013-10-07 (Actual)

PRIMARY OUTCOMES:
To determine the safety, tolerability, and recommended phase II dosing regimen of each GSK1120212-based treatment combination | Duration of study (approximately 3 years)

SECONDARY OUTCOMES:
To characterize population pharmacokinetic parameters | Duration of study (approximately 3 years)
To evaluate the anti-tumor activity as assessed by tumor response rate according to RECIST v1.1 | Duration of study (approximately 3 years)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (19):
- United States (13):
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Duarte, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Tyler, Texas
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Vancouver, Washington
- GSK Investigational Site, Toronto, Ontario, Canada
- France (4):
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Saint-Herblain
  - GSK Investigational Site, Toulouse
- GSK Investigational Site, Seoul, South Korea

REFERENCES:
- [Derived] Gandara DR, Leighl N, Delord JP, Barlesi F, Bennouna J, Zalcman G, Infante JR, Reckamp KL, Kelly K, Shepherd FA, Mazieres J, Janku F, Gardner OS, Mookerjee B, Wu Y, Cox DS, Schramek D, Peddareddigari V, Liu Y, D'Amelio AM Jr, Blumenschein G Jr. A Phase 1/1b Study Evaluating Trametinib Plus Docetaxel or Pemetrexed in Patients With Advanced Non-Small Cell Lung Cancer. J Thorac Oncol. 2017 Mar;12(3):556-566. doi: 10.1016/j.jtho.2016.11.2218. Epub 2016 Nov 19. PMID 27876675
- See also: Results for study 113486 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/113486?search=study&search_terms=113486#rs